CLINICAL TRIAL: NCT05595889
Title: Efficacy and Safety of Surufatinib Combined With Irinotecan as a Second-line Treatment for Small Cell Lung Cancer: a Single-arm, Prospective, Exploratory Clinical Study
Brief Title: Surufatinib Combined With Irinotecan as a Second-line Treatment for Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-E1-SCLC-001
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Small Cell Lung Cancer; Angiogenesis; Chemotherapy Effect
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — surufatinib; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib combined with irinotecan (Experimental): Surufatinib combined with irinotecan as a second-line treatment for small cell lung cancer
  Interventions: Drug: Surufatinib; Drug: Irinotecan

INTERVENTIONS:
Drug: Surufatinib — 250 mg/day p.o. QD
  Other Names: SULANDA
Drug: Irinotecan — Participants will receive irinotecan，100 mg/m2，Intravenous drip, day 1 and day 8 of every 3 weeks

SUMMARY:
To evaluate the clinical efficacy and safety of surufatinib combined with irinotecan in the second line treatment of small cell lung cancer.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, 40 patients with small cell lung cancer who failed to receive standard first-line therapy were selected to evaluate the efficacy and safety of surufatinib combined with irinotecan in the second-line treatment of small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years; Volunteer to participate in the trial and sign informed consent;
* Small cell lung cancer diagnosed by histopathology;
* Previous failure to receive first-line standard treatment was defined as intolerable toxic and side effects, disease progression during treatment, or recurrence after treatment; Intolerability was defined as grade IV (thrombocytopenia grade III and above) for hematologic toxicity and grade III or above for nonhematologic toxicity. Note: Each line of drug refers to medication for at least 1 cycle regardless of single drug or multi-drug combination;
* ECOG score: 0-1;
* At least one lesion detectable by CT, according to RECIST 1.1;
* Expected survival ≥12 weeks;
* At least one measurable lesion (RECIST 1.1 criteria, see Appendix 2);
* The functions of major organs and bone marrow are basically normal:
* Blood routine: white blood cell ≥ 4.0 x 109/L, neutrophil ≥ 1.5 x 109/L, platelet ≥ 100 x 109/L, hemoglobin ≥ 90 g/L; A) International normalized ratio (INR) ≤1.5× upper limit of normal (ULN), and activated partial thromboplastin time (APTT) ≤1.5×ULN; B) Liver function: total bilirubin ≤ 1.5 x ULN; In the absence of liver metastasis, ALT/AST /ALP ≤ 2.5 x ULN; ALT/AST /ALP ≤ 5 x ULN in patients with liver metastasis; C) Renal function: serum creatinine ≤ 1.5 x ULN, and creatinine clearance (CCr) 60 mL/min (see Appendix 6); D) Normal cardiac function, left ventricular ejection fraction (LVEF) ≥ 50% by two-dimensional echocardiography.
* Brain metastases must have been asymptomatic or treated and stabilized after discontinuation of steroids and anticonvulsants for at least 1 month prior to study treatment;
* Patients of childbearing age (including female and female partners of male patients) must take effective birth control measures;
* Good compliance is expected, and the efficacy and adverse reactions can be followed up according to the protocol requirements.

Exclusion Criteria:

* Small cell lung cancer with other pathological types of tumors;
* Previously received anti-angiogenic drugs, including bevacizumab, sovanitinib, sunitinib, sorafenib, anlotinib, apatinib, etc.
* Receive the following treatments within the first 4 weeks of treatment, including but not limited to surgery, chemotherapy, radical radiotherapy, biotargeted therapy, immunotherapy, and other investigational drugs;
* Pregnant or lactating women;
* With pleural effusion or ascites, respiratory syndrome (≥CTC AE grade 2 dyspnea);
* Symptomatic brain or meningeal metastases (except those who have undergone local radiotherapy or surgery for brain metastases for more than 6 months and have stable disease control);
* Severe infection (e.g., intravenous infusion of antibiotics, antifungals, or antivirals) within 4 weeks prior to treatment, or unexplained fever > 38.5 ° C during screening/initial administration;
* Hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
* The urine routine indicated urinary protein ≥2+, and 24-hour urinary protein quantity >1.0g;
* Obvious clinical bleeding symptoms or obvious bleeding tendency within 3 months before treatment (bleeding > 30 mL within 3 months, hematemesis, melanism, blood in stool), hemoptysis (fresh blood > 5 mL within 4 weeks), etc. Or treatment for a venous/venous thrombotic event in the previous 6 months, such as a cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; Long-term anticoagulant therapy with warfarin or heparin or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day) is required;
* Active heart disease, including myocardial infarction and severe/unstable angina, developed 6 months before treatment. Echocardiography showed left ventricular ejection fraction < 50% and poor arrhythmia control (including QTcF interval, > 450 ms in men and > 470 ms in women).
* The patient had had other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) within the previous 3 years or at the same time.
* Known allergy to the study drug or any of its excipients;
* Active or uncontrolled severe infections;

  1. Known human immunodeficiency virus (HIV) infection;
  2. A known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must exclude active HBV infection, i.e., HBV DNA positivity (>1×104 copies /mL or >2000 IU/ mL);
  3. Known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, liver cirrhosis];
* Any other disease, with clinical significance of metabolic abnormalities, abnormal physical examination or laboratory abnormalities, according to researchers, there is reason to suspect the patient has not suitable for the use of study drugs of a disease or condition (such as have a seizure and require treatment), or will affect the interpretation of results, or to make patients in high-risk situations;
* Other conditions deemed inappropriate for inclusion by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS was defined as the time from randomization until the date of first occurrence of investigator-assessed radiological disease progression or death due to any cause, whichever came first.

SECONDARY OUTCOMES:
Objective remission rate (ORR) | up to 12 months
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and kept for a certain time, including cases of complete remission and partial remission.
Disease control rate | up to 12 months
  The percentage of patients with complete response, partial response, and stable disease for more than 4 weeks in whom response could be evaluated.
Overall survival（OS） | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  OS was defined as the time from the date of randomization to the date of death due to any cause. For subjects who were alive or lost to follow-up by the data analysis cut-off date, survival was censored at the subject's last known survival time.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong He, Study Chair — Fujian Cancer Hospital

IPD SHARING:
Plan to Share IPD: No